CLINICAL TRIAL: NCT06149663
Title: Expanded Access Treatment with LP352 for Patients with Developmental and Epileptic Encephalopathies (DEEs) Who Successfully Completed an LP352 Clinical Trial (Intermediate-Size EAP)
Brief Title: Intermediate-Size Expanded Access Protocol (EAP) for LP352
Status: Available | Type: Expanded Access
Sponsor: Longboard Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: LP352-EAP-01
Record Dates: First submitted 2023-11-19; First posted 2023-11-29 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-02

CONDITIONS: Dravet Syndrome; Lennox Gastaut Syndrome; Developmental and Epileptic Encephalopathies
Keywords: CDKL5 deficiency disorder; developmental and epileptic encephalopathy; Dravet Syndrome; epilepsy; Lennox Gastaut Syndrome; treatment resistant epilepsy; tuberous sclerosis complex
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome; CDKL5 deficiency disorder; Epilepsy; Tuberous Sclerosis

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: LP352 — LP352 will be administered as a liquid either orally or through a G-tube or Percutaneous Endoscopic Gastrotomy (PEG) tube.

SUMMARY:
This is an intermediate-size expanded access program (EAP) study. The purpose of this EAP is to provide continued access to LP352, an investigational drug product being investigated in participants with DEEs. The EAP study will allow continued treatment with LP352 for eligible participants diagnosed with treatment resistant DEEs who successfully completed an LP352 Clinical Trial (Enrollment by Invitation) or an immediate family member who has the exact same gene mutation resulting in the same DEE epilepsy syndrome phenotype or a patient who previously participated in the lorcaserin EAP.

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or participant's legally authorized representative is willing and able to provide a written informed consent or assent form before participation in this EAP. An assent should be obtained from the patient, if possible. Assent must be obtained for adolescent EAP patients (<18 years of age) as required by local regulations.
2. Participant with DEE who has successfully completed an LP352 Clinical Trial.
3. Participant currently has clinical benefit from LP352 treatment, as assessed by their Treating Physician.
4. Participant currently tolerates LP352 treatment and has no safety issue which would prevent continued treatment.

Exclusion Criteria:

1. Participant was discontinued from an LP352 Clinical Trial for any reason.
2. Any serious and/or unstable new medical condition, psychiatric disorder, or other conditions at the time of transition to this EAP that could interfere with patient's safety, obtaining informed consent, assent, or compliance to this EAP protocol, in the opinion of the Treating Physician.

Ages: 2 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (22):
- United States (19):
  - Rancho Research Institute, Downey, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of California Benioff Childrens Hospital, San Francisco, California
  - Colorados Childrens Hospital, Aurora, Colorado
  - Northwest Florida Clinical Research Group, Gulf Breeze, Florida
  - Research Institute of Orlando, Orlando, Florida
  - University of Southern Florida, Tampa, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Northwestern Medicine Feinberg School of Medicine, Chicago, Illinois
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Corewell Health, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - New York University (NYU), New York, New York
  - Lenox Hill Hospital, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Providence Brain & Spine, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Children's Neuro Consultants of Austin, Austin, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (3):
  - Austin Hospital, Heidelberg, Heidelberg, Melbourne
  - Alfred Hospital, Melbourne, Melbourne
  - Children's Health Queensland Hospital and Health Service,, South Brisbane, Queensland